CLINICAL TRIAL: NCT03050983
Title: Observational Investigation to Determine Clinical Impact of Continuous Surveillance Monitoring (SM) on General Care Floors With a Nested Study to Determine the Clinical Utility of IPI (Integrated Pulmonary Index).
Brief Title: Determination of the Clinical Impact of Continuous Surveillance Monitoring (SM) and Utility of IPI.
Acronym: IPI
Status: Completed | Type: Observational
Sponsor: Medtronic - MITG (Industry)
Responsible Party: Sponsor
Other Study IDs: COVMOPO0525
Record Dates: First submitted 2017-02-09; First posted 2017-02-13 (Actual); Last update posted 2020-09-30 (Actual); Status verified 2020-09

CONDITIONS: Respiratory Depression; Respiratory Insufficiency
Keywords: Respiratory Compromise
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (2):
- Phase I: Prospective observation of alarmed events on the general care floor with continuous capnography and pulse oximetry monitoring prior to enabling IPI.
- Phase II: Enable the Integrated Pulmonary Index (IPI) and IPI alarm for the prospective observation of alarmed events on the general care floor with continuous capnography and pulse oximetry monitoring.
  Interventions: Device: IPI

INTERVENTIONS:
Device: IPI — Enable the IPI algorithm and IPI alarm algorithm
  Other Names: Integrated Pulmonary Index (IPI)
  Groups: Phase II

SUMMARY:
Single site prospective observational nested study of bedside CS20p monitor on the GCF impeded into a retrospective review of the frequency of escalation of care with intermittent vitals signs compared to continuous respiratory monitoring.

DETAILED DESCRIPTION:
Single site observational study of alarms and workflow on the general care floor where continuous surveillance monitoring (SM) with capnography and pulse oximetry is the standard of care before and after the Integrated Pulmonary Index is enabled within the context of a historical review of frequency of escalation of care as a function of the frequency and method of monitoring respiratory status. Observation of alarms will be electronically recorded on a Clinical Observation Tool (COT or iPad) that will have a virtual view of the CS20p measurements and alarm alerts for 24 hours on several patients at the same time. Patients will only be enrolled for 24 hours of observation of alarm status with associated patient activity and clinical interventions. Observation data with IPI disabled prior to implementation of IPI/IPI alarms will be used to evaluate optimal alarm alert settings including an IPI alert when enabled. Observation will continue with IPI enabled and alarms adjusted to study clinical utility of IPI on the GCF.

ELIGIBILITY:
Inclusion Criteria:

1. Spontaneous breathing adults ≥ 18 years of age, both male and female
2. On dual parameter CS20p monitoring with both capnography and pulse oximetry per Vanderbilt standard of care to monitor patients for respiratory compromise.
3. Expected minimum duration of 24 hours of continued capnography and pulse oximetry monitoring.

Exclusion Criteria:

1. Those patients who are expected to be discharged within six hours on the randomly selected observation floor.
2. Those patients not on the randomly selected floor for observation.
3. Those subjects randomly removed from the selected floor for observation pool in order to limit the number of subjects to be observed.
4. Those subjects in rooms with limited Wi-Fi signal quality as per VUMC IT.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The target study population will be adult patients on the general care floors (GCF) units where the dual parameter CS20p monitor is installed and used according to the Vanderbilt University Medical Center (VUMC) standard of care. Only those patients monitored via the CS20p with both capnography and pulse oximetry (dual parameters) for standard of care may be enrolled for observation.
Sampling Method: Non-Probability Sample
Enrollment: 440 (Actual)
Dates: Start 2017-02-15 (Actual); Primary Completion 2018-01-26 (Actual); Study Completion 2020-09-10 (Actual)

PRIMARY OUTCOMES:
Clinical Utility of IPI and IPI Alarm | Not to exceed nine months of observation
  Adjusted Hospital Length of Stay in both Phases

SECONDARY OUTCOMES:
Clinical Impact of continuous surveillance capnography and pulse oximetry monitoring | Not to exceed 24 months of reported escalation of care events to the Principal Investigator
  Number of alarms per patient, number of rapid response team activation, number of intensive care unit escalation and hospital cost per patient in each Phase.

CONTACTS AND LOCATIONS:
Overall Officials: Liza Weavind, MBBCh,FCCM,MMHC, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No
No plan to share